CLINICAL TRIAL: NCT00756717
Title: A Pilot Study of MK-0752 in Combination With Tamoxifen or Letrozole in Patients With Early Stage Breast Cancer Prior to Surgery
Brief Title: Study Of MK-0752 In Combination With Tamoxifen Or Letrozole to Treat Early Stage Breast Cancer
Acronym: MK-0752
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Loyola University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Kathy Albain, Assistant Professor, Loyola University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 200431
Record Dates: First submitted 2008-09-19; First posted 2008-09-22 (Estimated); Results first posted 2019-09-04 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: Breast Cancer
Keywords: MK-0752; Tamoxifen; Letroxole
MeSH Terms: conditions — Breast Neoplasms | interventions — 3-(4-((4-chlorophenyl)sulfonyl)-4-(2,5-difluorophenyl)cyclohexyl)propanoic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MK-0752 (Experimental): Oral gamma-secretase inhibitor drug MK-0752, 350 mg for three days, four days off, then three days on, over a period of 10 days
  Interventions: Drug: MK-0752

INTERVENTIONS:
Drug: MK-0752 — Women who are post menopausal will receive letrozole 2.5 mg by mouth one time per day for 24 days. Women who are pre menopausal, or who have a contraindication to letrozole will receive tamoxifen 20 mg orally one time per day for a period of 24 days. Starting on day 15 of this 24 day period all patients will receive the oral gamma-secretase inhibitor drug MK-0752 at a dose of 350 mg for three days on, then off four days, then three days on, for a total of 6 doses over a period of 10 days.

SUMMARY:
The purpose of this research project is to study the effect of a research (investigational) drug, MK-0752 combined with either tamoxifen or letrozole on breast cancer cells.

Tamoxifen and letrozole are standard hormone treatments used to treat breast cancers that are positive for the estrogen receptor. However, over time the breast cancer cells can become resistant to tamoxifen and letrozole. MK-0752 is in a class of drugs called gamma secretase inhibitors. Gamma secretase inhibitors may play a role in reversing the resistance to drugs such as tamoxifen and letrozole.

DETAILED DESCRIPTION:
OBJECTIVES

To evaluate the safety and tolerability of the gamma-secretase inhibitor MK-0752 in the pre-surgical setting in patients with early stage, estrogen receptor (ER) positive breast cancer, in combination with tamoxifen or an aromatase inhibitor (AI).

To establish the feasibility and success of multi-laboratory collaborations in evaluating clinical specimens and biomarker testing.

To provide preliminary data on the impact of MK-0752 on a panel of biomarkers involved in the notch signaling pathway.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed early stage, ER-positive (Allred score ≥3), invasive breast cancer that is not either locally advanced by criteria other than size or inflammatory, and is not metastatic. - Patients must be candidates for surgical removal of the tumor by lumpectomy or mastectomy.
* Patients must not have bilateral tumors. Tumor must be amenable to core biopsy in midstudy.
* Patients must be >18 years of age.
* Patients must have a performance status ≤1 by Zubrod criteria.
* Patients must have a life expectancy of greater than three months.
* Patients must have normal organ and marrow function within 28 days of registration as defined below:

  * absolute neutrophil count >1,500/μL
  * platelets >100,000/μL
  * total bilirubin ≤1.5 x the institutional upper limit of normal
  * AST(SGOT)/ALT(SGPT) <2 X institutional upper limit of normal
  * creatinine within normal institutional limits OR
  * creatinine clearance >60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
* Women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. A negative serum pregnancy test must be obtained within 72 hours of receiving the first dose of the hormonal therapy as well as within 72 hours of the first dose of the MK-0752 GSI medication for women of child-bearing potential. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

Exclusion Criteria:

* Patients may not have received any prior chemotherapy or endocrine therapy (tamoxifen, raloxifene, or an aromatase inhibitor) and may not have received prior therapy with a gamma-secretase inhibitor or other investigational agents. - Patients may not have received previous radiation therapy.
* Patients may not be currently participating or have participated in a study with an investigational compound or device within 30 days.
* Patients must not have known brain or CNS disease, evidence of brain or CNS metastases, or carcinomatous meningitis.
* Patients must not have an uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients may not have known hypersensitivity to the components of MK-0752 or it analogs.
* Patients will be excluded if there is a known history of human immunodeficiency (HIV) virus infection, or a known history of hepatitis B or C infection.
* Patients must not have a previous history of inflammatory bowel disease or uncontrolled irritable bowel syndrome.
* Patients must not have a history of greater than one basal cell carcinoma of the skin within the past five years or a history of Gorlin syndrome.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-02-14 (Actual); Primary Completion 2011-12-21 (Actual); Study Completion 2011-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Albain, MD, Principal Investigator — Loyola University
Locations (1):
- Loyola Univeristy Medical Center, Cardinal Bernardin Cancer Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers

REFERENCES:
- [Derived] Tabares-Seisdedos R, Rubenstein JL. Inverse cancer comorbidity: a serendipitous opportunity to gain insight into CNS disorders. Nat Rev Neurosci. 2013 Apr;14(4):293-304. doi: 10.1038/nrn3464. PMID 23511909

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MK-0752
Started | 22
Completed | 20
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: The baseline analysis population comprises the participants who completed the trial.
Arm/Group | MK-0752
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing at Least One Adverse Event
Description: The number of participants experiencing at least one adverse event during the 24-day observation period and initial post-operative visit.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | MK-0752
Number analyzed (Participants) | 20
Participants
  At least one adverse event | 15
  No Adverse Events | 5

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 30 days
Arm/Group | MK-0752
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 15/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-0752 (N=20)
Mild hot flashes (General disorders) | 8 (8)
Grade 1 Pelvic heaviness & vaginal discharge (General disorders) | 1 (1)
Grade 1 peri-orbital edema and cough (General disorders) | 1 (1)
Grade 1 acneiform facial rash (General disorders) | 4 (4)
Self-limiting nausea, vomiting, and headaches (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
There are no limitations or caveats to report.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes